CLINICAL TRIAL: NCT02374788
Title: Health Promotion in the Primary Care Setting- an Evaluation of the Sophia Step Study- a Structured Behaviour Change Program Focusing on Physical Activity in Persons With Pre- and Type 2 Diabetes
Brief Title: Sophia Step Study - a Behaviour Change Program on Physical Activity in Persons With Pre- and Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sophiahemmet University (Other)
Collaborators: Karolinska Institutet (Other); Uppsala University (Other); Arizona State University (Other)
Responsible Party: Principal Investigator, Unn-Britt Johansson, Unn-Britt Johansson, Sophiahemmet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SophiahemmetU
Record Dates: First submitted 2015-01-28; First posted 2015-03-02 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Type 2 Diabetes; Prediabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Participants in the intensive intervention group (A) receive a pedometer intervention and 12 group meetings over two years' time, with the majority of meetings being held in the first 6 months. The group meetings constitutes of a 30 min walk and 60 min group consulting based on techniques for behaviour change using an interactive program with positive feed-back following their steps on a website. One occasion is taking place at a gym with instruction for a home-based strength training program. Participants receive 10 individual consultations with a diabetes specialist nurse.
  Interventions: Behavioral: Pedometer intervention; Behavioral: Group meetings; Behavioral: Individual consultations
- Group B (Experimental): Participants in the pedometer group (B) receive a pedometer intervention. Henceforth they are left to continue by they own for two years.
  Interventions: Behavioral: Pedometer intervention
- Group C (No Intervention): The control group (C) receive diabetes care as usual except for the extra measurements included in the study. Diabetes care as usual is meeting a diabetes specialist nurse and a general practitioner once a year receiving lifestyle advice and physical activity on prescription.

INTERVENTIONS:
Behavioral: Pedometer intervention — Intensive intervention with pedometer. The participants are instructed to set daily step goal and to record their daily steps on a website.
  Arms: Group A; Group B
Behavioral: Group meetings — Participants receive 12 group meetings over two years' time.
  Arms: Group A
Behavioral: Individual consultations — Participants receive 10 individual meetings with a diabetes specialist nurse. Physical activity on prescription is used to set individual goals and to highlight the importance of physical activity.
  Arms: Group A

SUMMARY:
The aim of the study is to investigate the effects of two levels of primary care physical activity interventions on metabolic control and cardiovascular risk factors, compared to usual care in patients with pre- and type 2 diabetes.

The hypothesis is that both levels of interventions have effect on HbA1c with the more intense Group intervention having superior effects.

DETAILED DESCRIPTION:
Regularly physical activity may decrease the risk for type 2 diabetes, cardiovascular diseases, overweight and premature deaths. Despite the evidence that physical activity is beneficial to health,it is often ignored and underused aspect in diabetes care. The aim of the study is to investigate the effects of two levels of primary care physical activity interventions on metabolic control and cardiovascular risk factors, compared to usual care in patients with pre- and type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

Ability to communicate in Swedish Age 40-80 years Type 2 diabetes: Diagnosed type 2 diabetes with a duration of >=1 year Pre-diabetes: HbA1c >39-<47, Fasting plasma glucose >5.6 mmol/l

Exclusion Criteria:

* Myocardial infarction in the past 6 months
* serum creatinine >140
* diabetic ulcer or risk for ulcer
* prescribed insulin in past 6 months
* additional disease prohibiting physical activity
* have experienced repeated hypoglycaemia or severe hypoglycaemia in past 12 months
* classified in very hard-intensity activity according to Stanford Brief Activity Survey
* having no access to internet.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2013-11; Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

PRIMARY OUTCOMES:
HbA1c (mmol/mol) | up to month 24.
  Haemoglobin A1c

SECONDARY OUTCOMES:
fasting plasma glucose (mmol/L) | week 0, 12, 24, and month 9, 12, 18 and 24.
  Determined by a glucose oxidase method
Physical activity level (counts/min) | week 0 and month 6, 12, 18, 24
  Actigraph accelerometer GT1M
Steps/day | week 0, 8, 12, 16, 24, and month 9, 12, 18 and 24.
  Actigraph accelerometer GT1M
fasting-Insulin (mU/l) | week 0, 12, 24, and month 12 and 24.
  Serum insulin concentrations are determined with RIA-kits purchased from Pharmacia & Upjohn, Stockholm.
LDL (mmol/L) | week 0, 12, 24, and month 12 and 24.
  LDL is determined by using a homogeneous method (lowdensity lipoprotein)
Total cholesterol (mmol/L) | week 0, 12, 24, and month 12 and 24.
  total Cholesterol is determined by using enzymatic method
IGF BP1 (μg/L) | week 0, 12, 24, and month 12 and 24.
  insulin-like growth factor binding protein 1
Free fatty acids (mmol(L ) | week 0, 12, 24, and month 12 and 24.
  Samples are saved for later free fatty acid analyses.
Triglycerides (mmol/L) | week 0, 12, 24, and month 12, 18 and 24.
  Triglycerides is determined by using enzymatic method (Triglycerides)
HDL (mmol/L) | week 0, 12, 24, and month 12, 18 and 24.
  HDL is determined by using a homogeneous method (lowdensity lipoprotein)(High-density lipoprotein)
ApoB (g/l) | week 0, 24 and month 24.
  Apolipoprotein B is determined by using turbimetric method
ApoA1 (g/l) | week 0, 24 and month 24.
  ApolipoproteinA1 is determined by using turbimetric method
C-peptide (pmol/l) | week 0, 12, 24, and month 12 and 24.
  C-peptid are determined by using immunometric method using two monoclonal antibodies and detection with electrochemiluminiscense using a Modular E system (Beckman Coulter, Inc.).
BMI (kg/m2) | week 0,8, 12,16, 24, and month 9, 12, 18 and 24.
  Body mass index
Weight (kg) | week 0,8, 12,16, 24, and month 9, 12, 18 and 24.
  Tanita digital scale (Model TBF- 300A, Arlington Heights, IL). Weight is measured with light clothes, no shoes to the nearest 0.1 kg.
% Body Fat | week 0,8, 12,16, 24, and month 9, 12, 18 and 24.
  % Body Fat is determined by Tanita digital scale (Model TBF- 300A, Arlington Heights, IL).
Waist circumference (cm) | week 0,8, 12,16, 24, and month 9, 12, 18 and 24.
  Waist circumference is measured with SECA 201 tape, horizontal around the waist 2 cm above the umbilicus.
Sagittal Abdominal Diameter (cm) | week 0,8, 12,16, 24, and month 9, 12, 18 and 24.
  Sagittal abdominal diameter is measured with the subject in a supine position with the knees expanded at the level of the umbilicus using a Holtain-Kahn abdominal caliper (Holtain, Ltd., Crosswell, Crymych; Dyfed, UK).
Resting blood pressure (mmHg) | week 0,8, 12,16, 24, and month 9, 12, 18 and 24.
  diastolic blood pressure and systolic blood pressure. Resting blood pressure is measured with Omron M6 Comfort.
Muscle strength | week 0, 12, 24, and month 9, 12, 18 and 24.
  measured by hand-held dynamometry. Hand grip strength is measured in kilograms using the hand-held Saehan Hydraulic Hand Dynamometer, model SH5001 (former Jamar) (Saehan Corporation, Masan, South Korea).
Change in Smoking and snuffing habits | Evaluation is conducted at baseline and at 24 months after completion of the intervention period
  Change in Smoking and snuffing habits is measured with questions on current and previous habits and the dose

OTHER OUTCOMES:
Change in Dietary habits | Evaluation is conducted at baseline and at week 8, 12, 24 and month 12 and 24 after completion of the intervention period
  Change in Dietary habits is measured by a set of questions developed and validated by The Swedish National Food Agency.
Change in Alcohol habits | Evaluation is conducted at baseline and at week 24 and month 12 and 24 after completion of the intervention period
  Change in Alcohol habits is measured by two questions from AUDIT-The alcohol Use disorders
Change in Stress and working condition | Evaluation is conducted at baseline and at week 12, 24 and month 12 and 24 after completion of the intervention period
  Change in Stress and working condition is measured by four questions
EuroQol (EQ-5D) | week 0, 12, 24 and month 12 and 24
  measured by EQ-5D assess components of health related QoL (HRQoL). EQ-5D includes measures related to mobility, hygiene, daily activities, pain/ discomfort and anxiety/depression.
Sleep | Evaluation is conducted at baseline and at week 12, 24 and month 12 and 24 after completion of the intervention period
  Sleep is measured by two questions. One question on difficulties falling asleep and one question on sleep quality.
Self reported physical activity | week 0, 12, 24 and month 12 and 24
  International Physical Activity Questionnaire (IPAQ) self-reported 7-item questionnaire to assess physical activity.
Self-efficacy for exercise | week 0, 12, 24 and month 12 and 24
  The questionnaire Self-efficacy for exercise is a 5 item questionnaire and assess one´s confidence to continue exercising in different situations.
Physical Activity Social Support (PASS) | week 0, 12, 24 and month 12 and 24
  Physical Activity Social Support (PASS) for exercise 6 items.
Change in Neighborhood Environment | Evaluation is conducted at baseline and at week 12, 24 and month 12 and 24 after completion of the intervention period
  Change in Neighborhood Environment is measured by 17 questions about Walking Environment, Availability of healthy Foods, Safety and Social cohesion
Change in Perceived Stress Scale (PSS) | Evaluation is conducted at baseline and at week 12, 24 and month 12 and 24 after completion of the intervention period
  Change in Perceived Stress is measured by the Perceived Stress Scale (PSS) which is a 14- items questionnaire.
Change in diabetes distress (PAID-20) | Evaluation is conducted at baseline and at week 12, 24 and month 12 and 24 after completion of the intervention period
  Diabetes distress is measured by The Problem Areas in Diabetes questionnaire (Swe-PAID-20): This is a 20 items questionnaire
Hospital Anxiety and Depression Scale (HADS) | week 0, 12, 24 and month 12 and 24
  HADS is a 14 item questionnaire and consists of two subscales depression and anxiety, with seven items each.

CONTACTS AND LOCATIONS:
Overall Officials: Unn-Britt Johansson, Professor, Principal Investigator — Sophiahemmet University
Locations (1):
- Sophiahemmet University, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossen J, Yngve A, Hagstromer M, Brismar K, Ainsworth BE, Iskull C, Moller P, Johansson UB. Physical activity promotion in the primary care setting in pre- and type 2 diabetes - the Sophia step study, an RCT. BMC Public Health. 2015 Jul 12;15:647. doi: 10.1186/s12889-015-1941-9. PMID 26164092
- [Derived] Larsson K, Von Rosen P, Rossen J, Johansson UB, Hagstromer M. Relative time in physical activity and sedentary behaviour across a 2-year pedometer-based intervention in people with prediabetes or type 2 diabetes: a secondary analysis of a randomised controlled trial. J Act Sedentary Sleep Behav. 2023 Jun 1;2(1):10. doi: 10.1186/s44167-023-00020-w. PMID 40217375
- [Derived] Larsson K, Rossen J, Norman A, Johansson UB, Hagstromer M. Predictors associated with an increase in daily steps among people with prediabetes or type 2 diabetes participating in a two-year pedometer intervention. BMC Public Health. 2024 May 11;24(1):1290. doi: 10.1186/s12889-024-18766-6. PMID 38734659
- [Derived] Rossen J, Larsson K, Hagstromer M, Yngve A, Brismar K, Ainsworth B, Aberg L, Johansson UB. Effects of a three-armed randomised controlled trial using self-monitoring of daily steps with and without counselling in prediabetes and type 2 diabetes-the Sophia Step Study. Int J Behav Nutr Phys Act. 2021 Sep 8;18(1):121. doi: 10.1186/s12966-021-01193-w. PMID 34496859
- [Derived] Rossen J, Hagstromer M, Yngve A, Brismar K, Ainsworth B, Johansson UB. Process evaluation of the Sophia Step Study- a primary care based three-armed randomized controlled trial using self-monitoring of steps with and without counseling in prediabetes and type 2 diabetes. BMC Public Health. 2021 Jun 22;21(1):1191. doi: 10.1186/s12889-021-11222-9. PMID 34157994
- [Derived] Rossen J, Von Rosen P, Johansson UB, Brismar K, Hagstromer M. Associations of physical activity and sedentary behavior with cardiometabolic biomarkers in prediabetes and type 2 diabetes: a compositional data analysis. Phys Sportsmed. 2020 May;48(2):222-228. doi: 10.1080/00913847.2019.1684811. Epub 2019 Nov 12. PMID 31663410
- See also: Study protocol — http://bmcpublichealth.biomedcentral.com/articles/10.1186/s12889-015-1941-9